CLINICAL TRIAL: NCT03840421
Title: GP Vs PF As Induction Chemotherapy Combined with CCRT for Locoregionally Advanced Nasopharyngeal Carcinoma：a Prospective,Parallel, Randomized, Open Labeled, Multicenter Phase III Clinical Trial
Brief Title: GP Vs PF As Induction Chemotherapy Combined with CCRT for Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital, China (Unknown); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-140
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nasopharyngeal Diseases; Head and Neck Neoplasm
Keywords: gemcitabine; cisplatin; fluorouracil
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nasopharyngeal Diseases; Head and Neck Neoplasms | interventions — Gemcitabine; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- gemcitabine and cisplatin (Experimental): Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 2 cycles.
  Interventions: Drug: gemcitabine and cisplatin; Radiation: IMRT; Drug: cisplatin
- cisplatin and fluorouracil (Active Comparator): Patients receive fluorouracil (800mg/m² d1-5) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 2 cycles.
  Interventions: Drug: cisplatin and fluorouracil; Radiation: IMRT; Drug: cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin — Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before concurrent chemoradiotherapy.
  Other Names: gemcitabine and cisplatin (GP)
  Arms: gemcitabine and cisplatin
Drug: cisplatin and fluorouracil — Patients receive fluorouracil (800mg/m2 d1-5) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before concurrent chemoradiotherapy.
  Other Names: cisplatin and fluorouracil (PF)
  Arms: cisplatin and fluorouracil
Radiation: IMRT — Intensity modulated-radiotherapy (IMRT) is given as 30～33 fraction with five daily fractions per week for 6-7 weeks to a total dose of 68～70 Gy to the primary tumor
Drug: cisplatin — IMRT concurrently with cisplatin 100 mg/m² every 3 weeks for 2 cycles.
  Other Names: cisplatin（DDP）

SUMMARY:
The purpose of this study is to compare the survival and toxicity of GP (gemcitabine and cisplatin) vs. PF (cisplatin and fluorouracil) as induction chemotherapy combined with concurrent chemoradiotherapy (CCRT) for locoregionally advanced nasopharyngeal carcinoma( NPC ) patients.

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage T1-4N2-3/T4N0-1M0 are randomly assigned to receive GP (gemcitabine and cisplatin) or PF (cisplatin and fluorouracil) induction chemotherapy combined with concurrent chemoradiotherapy. Patients in both arms receive radical radiotherapy, and cisplatin (100mg/m²) every three weeks for two cycles during radiotherapy. Patients in the investigational arm receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for three cycles. Patients in the control arm receive fluorouracil (800mg/m² d1-5) and cisplatin (80mg/m² d1) every 3 weeks for three cycles. Our primary endpoint is progress-free survival (PFS). Secondary end points include distant metastasis-free survival (DMFS), overall survival (OS), locoregional relapse-free survival (LRRFS), initial response rates after treatments, toxic effects and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Tumor staged as T1-4N2-3/T4N0-1M0（according to the 8th AJCC edition）
* Male and no pregnant female
* Age between 18-65
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <2.0×upper limit of normal (ULN)
* Adequate renal function: creatinine clearance ≥60 ml/min
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70
* Without radiotherapy or chemotherapy
* Patients must give signed informed consent

Exclusion Criteria:

* Evidence of relapse or distant metastasis
* History of prior malignancy or previous treatment for NPC
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
progress-free survival (PFS) | 3 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site.

SECONDARY OUTCOMES:
Distant Metastasis-Free Survival (DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Overall Survival (OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Number of participants with adverse events | up to 3 years
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China